CLINICAL TRIAL: NCT04142723
Title: Alcoholic Hepatitis in Latin-America: A Prospective and Multicentric Study (AH-LATIN).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: ALEH (Unknown); Hospital Nacional Hipolito (Unknown); Hospital Goyoneche Arequipa (Unknown); Hospital Nacional Edgardo Rebagliati Martins (Other); HBCASE (Unknown); Hospital Regional Honorio Delgado Arequipa Peru (Unknown); Hospital Nacional Daniel Alcides Carrión - Callao (Unknown); Instituto de Gastroenterología (Unknown); Hospital Docente Clinico Quirurgico:Manuel Piti Fajardo (Unknown); Hospital de Clínicas D. N. Avellaneda (Unknown); Hospital Padilla. Tucuman (Unknown); Hospital Pablo Soria. Jujuy (Unknown); FUNDACIÓN SAYANI (Unknown); Hospital Italiano Buenos Aires (Unknown); Rosario (Unknown); Hospital de Gastroenterología Dr Carlos Bonorino Udaondo (Unknown); Hospital Austral de Buenos Aires (Unknown); Francisco Alfonso Solís Galindo (Unknown); Centro de Investigación en Enfermedades Hepáticas y Gastroenterología (Unknown); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Hospital General de Mexico (Other Government); Hospital Eugenio Espejo (Unknown); Hospital de Especialidades de las FF.AA Quito (Unknown); Hospital Carlos Andrade Marín (Unknown); Hospital General San Juan de Dios (Unknown); Hospital Roosevelt (Unknown); Hospital San Vicente Fundación Medellín (Unknown); Clinica Universitaria Colombia (Unknown); Hospital San Vicente Fundación - Rionegro (Unknown); Fundacion Cardioinfantil (Unknown); Hospital Pablo Tobon Uribe. Univ. De Antioquia (Unknown); Fundação Hospital Adriano Jorge (Unknown); Hospital do Rocio (Unknown); Hospital das Clinacas Riberao Preto (Unknown); Universidade Estadual Paulista (UNESP) - Botucatu/São Paulo (Unknown); FUNDHACRE- Serviço de Assistência Especializada- Acre (Unknown); Hospital Getúlio Vargas - Teresina/Piauí (Unknown); Hospital do Servidor Público Estadual - São Paulo/São Paulo (Unknown); Hospital Federal de Bonsucesso - Rio de Janeiro/Rio de Janeiro (Unknown); CHP/ Cl Davila / HCUH (Unknown); Hospital San Juan de Dios (Unknown); Hospital Sotero Del Rio (Unknown); Hospital San Borja-Arriaran (Other); University of Chile (Other); Hospital Clinico Universidad Catolica (Unknown); Hospital de Concepcion (Unknown); Hospital Escuela (Unknown)
Responsible Party: Sponsor
Other Study IDs: Alcoholic Hepatitis
Record Dates: First submitted 2019-10-02; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis, Alcoholic
Keywords: alcoholic, liver disease, cirrhosis
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood withdraw — venous blood sampling

SUMMARY:
The primary objective of this study is to determine the prevalence of AH in addition to its clinical characteristics and in-hospital mortality of patients that are hospitalized for AH in different hospitals across Latin American countries This study is carried out in different health centers throughout America, with all the countries belonging to the Latin American Association for the study of liver diseases (ALEH) more Canada and United States This would allow us to better understand the epidemiology of AH in our region and thus implement prevention measures with more solid data. Importantly, this would allow us to optimize therapeutic measures

DETAILED DESCRIPTION:
This study is sponsored and organized by the "group Latin American of interest special in the study of the disease hepatic Alcohol" (ALEH-GLEHA), belonging to the Latin American Association for the study of the hepatic illnesses (ALEH), which is an association non-profit that has nearly 1,000 members from most of the countries of Latin America.

All patients admitted to the hospital with suspected alcoholic hepatitis will be evaluated to see if they can be included in the study. Patients will be enrolled according with the inclusion and exclusion criteria.

The investigators will take a blood sample to be analyzed as part of the necessary data record, for the study of genes and identification of proteins involved in the development, evolution and prognosis of alcoholic hepatitis.

If the medical doctor had instructed to perform a liver biopsy, voluntarily the investigators will ask to participants donate a small share of the surplus of histological sample To achieve this, it is necessary to generate a data bank of clinical information and biological samples (blood, urine, bile, stools, salivary sample or tissue samples) that allows studying the various factors involved in the development and prognosis of this disease in the countries of the Americas.

The investigators will make a clinical follow-up for a year, consisting of phone calls to complete a questionnaire about participant's health. These calls will be made in month 1, 3, 6 and 12 subsequent to participant's hospital discharge.

The data collected are identified by a code and only the study physicians can correlate the data with the participants and medical history, so the participant's identity will not be shared.

There is no financial compensation associated with the study

ELIGIBILITY:
Inclusion Criteria:

1. Consumption of more than 3 drinks per day (40 g) in women and more than 4 drinks per day (50-60 g) in men.
2. Excessive alcohol consumption for more than 5 years in a row or interrupted.
3. No more than 60 days of abstinence before the onset of jaundice.
4. Bilirubin levels > 3 mg / dL (> 50 μmol / L), AST> 50 IU / mL, AST / ALT ratio> 1.5.
5. Absence of other causes of hepatic disease.

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy or lactation
3. Alcohol abstinence for more than 60 days before the event that led to hospitalization.
4. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels beyond 400 IU/ml.
5. Presence of drug-induced liver injury (DILI), ischemic hepatitis, biliary duct obstruction, viral hepatitis, autoimmune hepatitis or Wilson's disease.
6. Hepatocellular carcinoma beyond the Milan criteria (ie, a single lesion < 5 cm or no more than 3 lesions, the largest of which measures ≤ 3 cm).
7. Extrahepatic neoplasia with a life expectancy of less than 6 months.
8. History of severe extrahepatic disease (eg, chronic kidney failure requiring hemodialysis, severe heart disease (NYHA class ≥ 3), severe chronic lung disease that confers a survival of less than 6 months.
9. Patients who cannot provide informed consent and that lack a responsible legal substitute.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consumption of more than 3 drinks per day in women and more than 4 drinks per day in men
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of subjects hospitalized with alcoholic hepatitis who die at 30, 60 and 90 days. | 90 days
  To determine the clinical characteristics, complications and in-hospital mortality of patients who are hospitalized for alcoholic hepatitis in different establishments in America.
  To achieve this, it is necessary to generate a data bank of clinical information and biological samples (blood, urine, bile, stools, salivary sample or tissue samples) that allows studying the various factors involved in the development and prognosis of this disease in the countries of the Americas. This will help us to know aspects of the highest prevalence and mortality from alcoholic hepatitis in Latin Americans in comparison to other regions of the world and useful information in the prevention and early diagnosis of this disease.

SECONDARY OUTCOMES:
Number of subjects hospitalized with alcoholic hepatitis who develop complications (infection, gastrointestinal bleeding, renal failure, etc.) | 4 years
  Inquire about the incidence of infections and prevalence of infections resistant to antibiotics in patients hospitalized for alcoholic hepatitis.
Number of subjects with alcoholic hepatitis who are cataloged as responders by Lille score. | 4 years
  with the data bank researches will be able to track patients through health questionnaires
Mean Model of End-Stage Liver Disease (MELD) score at day 0, 30, 60 and 90. | 4 years
  with the data bank researches will be able to track patients through health questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: juan pablo p arab, md, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Unversidad Catolica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided